CLINICAL TRIAL: NCT06006377
Title: Investigation of the Efficacy of Treatments With Backup Device in Spine Pathologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar56
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Spine Disease; Back Pain; Disc Herniation
Keywords: Backup; physiotherapy
MeSH Terms: conditions — Spinal Diseases; Back Pain; Intervertebral Disc Displacement | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: conventional physiotherapy and backup device therapy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electrotherapy (Active Comparator): conventional physiotherapy methods (hotpack, Ultrasound , Transcutaneous Electrical Nerve Stimulation)
  Interventions: Other: electrotherapy
- backup (Experimental): conventional physiotherapy and backup device therapy
  Interventions: Other: Backup therapy

INTERVENTIONS:
Other: electrotherapy — hotpack electrotherapy ultrasound exercises
  Arms: electrotherapy
Other: Backup therapy — The backup spine health device is in the form of a mat and provides segmental electrical stimulation to the spines. At the same time, the mat can heat up to 40 degrees during the treatment process. Backup spine health device is very effective in both reducing pain and strengthening the muscles with electrical stimulations by reaching even the deep muscles around the spine. Sessions consist of 30 minutes
  Arms: backup

SUMMARY:
Our aim in this study is to examine the effectiveness of the Backup spine health device in spinal problems and compare it with traditional physical therapy methods.

DETAILED DESCRIPTION:
The investigators study was planned as a randomized controlled study. Participants will be divided into 2 groups as conventional physiotherapy and Backup group by simple randomized method. Participants will be taken to a treatment program for 12 weeks, 3 days a week. Parameters such as pain, posture, sleep quality, quality of life, muscle shortening at the beginning and end of the study. The results will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20-60
* sick individuals with spinal problems
* Persons who have filled out the consent form

Exclusion Criteria:

* People with spinal pathology for whom physiotherapy is contraindicated
* Having a neurological problem

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 14 weeks
  It is a 19-item self-report scale that evaluates sleep quality and impairment over the past month. It consists of 24 questions, 19 questions are self-report questions, 5 questions are questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleeping Drug Use, and Daytime Dysfunction. Each component is evaluated over 0-3 points. The total score of the 7 components gives the scale total score. The total score ranges from 0 to 21. A total score greater than 5 indicates "poor sleep quality".
World Health Organization Quality of Life Scale Short Form | 14 weeks
  The scale is a 26-item scale. Each section and area receives a maximum score of 20 points or 100 points. A high score indicates good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Asiye ÖNELGE, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lurie J, Tomkins-Lane C. Management of lumbar spinal stenosis. BMJ. 2016 Jan 4;352:h6234. doi: 10.1136/bmj.h6234. PMID 26727925
- [Background] Stoll T, Germann D, Hagmann H. [Physiotherapy in lumbar disc herniation ]. Ther Umsch. 2001 Aug;58(8):487-92. doi: 10.1024/0040-5930.58.8.487. German. PMID 11552355
- [Background] Andersen MO, Andresen AK, Lorenzen MD, Isenberg-Jorgensen A, Stottrup C. [Non-surgical treatment of lumbar radiculopathy]. Ugeskr Laeger. 2017 Nov 13;179(23):V05170397. Danish. PMID 29139353